CLINICAL TRIAL: NCT03491202
Title: The Genetic Basis for Atrial Fibrillation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jesse Brown VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Katherine Durham MS, APN, Cardiology Nurse Practitioner, Jesse Brown VA Medical Center
Other Study IDs: 977544
Record Dates: First submitted 2018-04-02; First posted 2018-04-09 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- atrial fibrillation: Patients with a diagnosis of atrial fibrillation will be eligible for enrollment

SUMMARY:
Atrial fibrillation (AF) is reaching epidemic proportions in the aging U.S. and European populations, but the mechanisms of increased susceptibility to atrial fibrillation are still unknown. In this study, we look to further examine genetic and medical co-morbidity influence of atrial fibrillation duration and response to medications. In Specific Aim 1, we propose the creation of a Veterans Affairs AF Biorepository (VAAFBio), which is a resource that will collect and store clinical, demographic, blood and DNA samples from patients with atrial fibrillation to aide this study and future studies of this type in the VA population. In Specific Aim 2, examine common genetic polymorphisms in veteran patients with atrial fibrillation and examine gene-environment interactions with risk factors for atrial fibrillation.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is reaching epidemic proportions in the aging U.S. and European populations, but the mechanisms of increased susceptibility to atrial fibrillation are still unknown. In this study, the investigators look to further examine genetic and medical co-morbidity influence of atrial fibrillation duration and response to medications. In Specific Aim 1, the investigators propose the creation of a Veterans Affairs AF Biorepository (VAAFBio), which is a resource that will collect and store clinical, demographic, blood and DNA samples from patients with atrial fibrillation to aide this study and future studies of this type in the VA population. In Specific Aim 2, the investigators will examine common genetic polymorphisms in veteran patients with atrial fibrillation and examine gene-environment interactions with risk factors for atrial fibrillation.

Patients will be identified through the VA inpatient and outpatient clinic, and will be approached for inclusion in the study. The target enrollment for the research and biorepository is 600 participants. A detailed family history, medical background, study questionnaires and a blood sample will then be obtained by the principal investigator or a research coordinator, following written informed consent under a protocol approved by the Jesse Brown VA Institutional Review Board. Once enough samples are collected, coded DNA samples will be sent out to analyze for linkage to known/candidate loci for AF.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18 years of age, and up to 100.
* Subjects must have a documented history of atrial fibrillation by ECG, ECHO, and or Holter monitor event recorder.
* Subjects must be willing to give written, informed consent.

Exclusion Criteria:

* Patients with a history of AF or atrial flutter that is only associated with cardiac surgery will be excluded from the study.
* Subjects who cannot speak English will be excluded from the study.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be identified in the outpatient clinic or in the inpatient setting at the Jesse Brown VA Medical Center and approached for informed consent and HIPAA authorization.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-05-25 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Symptoms related to atrial fibrillation (chest pain, dyspnea, palpitations) | 1 year
heart rate | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Jesse Brown VA Medical Center, Chicago, Illinois, United States